CLINICAL TRIAL: NCT05679505
Title: Effects of Vagus Nerve Stimulation in Post-COVID-19 Syndrome: A Randomized Controlled Trial
Brief Title: Vagus Nerve Stimulation for Post-COVID Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Alper Percin, Lecturer, Bahçeşehir University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY003
Record Dates: First submitted 2023-01-05; First posted 2023-01-11 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Long COVID; Vagus Nerve Stimulations; Heart Rates; Autonomic Nervous System Disorders
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Autonomic Nervous System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Left ear transcutaneous vagus nerve stimulation (Experimental): Left ear transcutaneous vagus nerve stimulation will be applied to the participants in this group.A continuous electrical stimulation with a current frequency of 10 Heartz (Hz) with a current transit time of 300 μs was applied to the participants in both groups. The participants included in both groups were treated with taVNS with the "Vagustim" device for 20 minutes once a day and for a total of 10 sessions application was made.
  Interventions: Device: Auricular transcutaneous vagus nerve stimulation
- Bilateral double ear transcutaneous vagus nerve stimulation (Experimental): Bilateral double ear transcutaneous vagus nerve stimulation will be applied to the participants in this group.A continuous electrical stimulation with a current frequency of 10 Heartz (Hz) with a current transit time of 300 μs was applied to the participants in both groups. The participants included in both groups were treated with taVNS with the "Vagustim" device for 20 minutes once a day and for a total of 10 sessions application was made.
  Interventions: Device: Auricular transcutaneous vagus nerve stimulation

INTERVENTIONS:
Device: Auricular transcutaneous vagus nerve stimulation — Transcutaneous vagus nerve stimulation (taVNS) was performed with an FDA-approved Vagustim stimulation device and an electrode-shaped earpiece. In the participants included in the study and randomized to two groups, i) left ear taVNS was applied to the first group and ii) double-ear taVNS was applied to the second group.

SUMMARY:
The aim of this study is to increase parasympathetic activity and decrease the severity of symptoms by providing vagal stimulation with the t-VNS method in order to suppress the increased sympathetic activity in patients with prolonged Covid symptoms.The main question[s] it aims to answer are:

Question 1:Is left ear transcutaneous vagus nerve stimulation effective in suppressing the symptoms of patients in Post Covid syndrome?

Question 2:Is bilateral auricular transcutaneous vagus nerve stimulation effective in suppressing the symptoms of patients in Post Covid syndrome?

A 5-minute heart rate variability measurement will be performed to measure the effectiveness of vagus nerve stimulation in participants.HRV is a non-invasive method used to evaluate ANS activity and is a measure of heart rate change over a period of time

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Experiencing at least one of the post-covid symptoms for 12 weeks or longer

Exclusion Criteria:

* Considering that the female reproductive hormones level in the body and menstrual cycle may affect the ANS in female patients, female participants in perimenopausal, post-menopausal and pregnancy conditions were excluded from the study.
* Participants who used medication for the treatment of ANS dysfunction in the last six months were also excluded from the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | After the evaluation of the patients on the first day of participation in the study, the final evaluation was completed at the end of the 10th session (10 days later).
  HRV is a non-invasive method used to evaluate ANS activity and is a measure of heart rate change over a period of time. It analyzes the change in the beat-beat intervals of the heart and reflects the balance between PNS and SNS. During the analysis of heart rate variability measurement, the results obtained from sub-parameters such as stress index, time-domain and frequency-domain measurements allow evaluation of PNS and SNS activity.

SECONDARY OUTCOMES:
Fatigue Severity Scale | After the evaluation of the patients on the first day of participation in the study, the final evaluation was completed at the end of the 10th session (10 days later).
  The Fatigue Severity Scale, which is applied in the form of a questionnaire to determine the severity of fatigue accompanied by chronic diseases, consists of a total of 9 questions and according to the results obtained, it gives results as No Fatigue (<2.8 points) and chronic fatigue syndrome (>6.1 points).

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Erenler, Prof. Dr., Study Chair — Igdir University
Locations (1):
- Iğdır State Hospital, Iğdır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No